CLINICAL TRIAL: NCT01109290
Title: Validation of Non-invasive Technologies for the Characterization of Sweat Gland Function in Patients With Recessively Inherited Hypohidrotic Ectodermal Dysplasia, Their Heterozygous Family Members and Healthy Controls
Brief Title: Characterization of Sweat Gland Function in Patients With Recessively Inherited Hypohidrotic Ectodermal Dysplasia
Status: Completed | Type: Observational
Sponsor: University Hospital Erlangen (Other)
Collaborators: Edimer Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Holm Schneider, Head of the Division of Molecular Pediatrics, University Hospital Erlangen
Other Study IDs: ED10
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Hypohidrotic Ectodermal Dysplasia
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- HED children
- HED adults
- Control children
- Control adults

SUMMARY:
Hypohidrotic ectodermal dysplasia (HED) is a complex genetic disorder characterized by lack of sweat glands, sparse hair, and missing or malformed teeth. Inability to sweat may result in episodes of severe hyperthermia and cause sudden infant death. To assess sweat gland function in HED patients, the investigators will first quantify gland pores in a defined area of the palm and then stimulate the glands by pilocarpine followed by sweat collection in a special capillary for volume determination. This will be combined with non-invasive skin conductance measurement prior and subsequent to stimulation of the sympathetic nervous system. The data should provide a basis for genotype-phenotype correlation.

ELIGIBILITY:
Inclusion Criteria:

* for patients: hypohidrotic ectodermal dysplasia caused by mutations in the genes EDA or EDAR
* written informed consent

Exclusion Criteria:

* febrile disease
* pregnancy or breastfeeding
* implantable electronic devices, e.g. pacemaker
* hypersensitivity to self-adhesive electrodes

Max Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: subjects with recessively inherited hypohidrotic ectodermal dysplasia (HED), their heterozygous family members and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holm Schneider, MD, Principal Investigator — University Hospital Erlangen
Locations (1):
- University Hospital Erlangen, Erlangen, Bavaria, Germany